CLINICAL TRIAL: NCT03290612
Title: Chronotherapeutic Use of Vitamin C to Reduce Morning Cardiovascular Risk
Brief Title: Vitamin C to Reduce Morning Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Steven A. Shea, Director, Oregon Institute of Occupational Health Sciences, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB 00017294
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Risk Factor
Keywords: Sleep; Vitamin C
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vitamin C and Placebo doses will be blinded by the research pharmacy, so that participants and investigators are masked to the identity of the tablet. Data analysis will be blinded to the conditions as well until the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C then Placebo (Experimental): Participants will receive a 1.5g dose of Ascorbic Acid upon wake for the first visit, and a placebo tablet on the second visit.
  Interventions: Dietary Supplement: Vitamin C; Other: Placebo
- Placebo then Vitamin C (Experimental): Participants will receive a placebo tablet upon wake for the first visit, and a 1.5g dose of Ascorbic Acid on the second visit.
  Interventions: Dietary Supplement: Vitamin C; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1.5g Ascorbic Acid
  Other Names: Ascorbic Acid
Other: Placebo — Inactive placebo to mimic 1.5g ascorbic acid.

SUMMARY:
This study will test the efficacy of Vitamin C to counteract morning cardiovascular (CV) risk markers in a randomized, double blind, placebo controlled crossover pilot study. The participants will also perform morning typical behaviors such as arousal from sleep, change in posture (getting out of bed) and mild intensity physical activity; identical to the stressors encountered in everyday life. Primary dependent variables are markers of cardiovascular risk including vascular endothelial function and oxidative stress.

DETAILED DESCRIPTION:
The investigators plan to test the efficacy of Vitamin C to counteract morning cardiovascular (CV) risk markers in a randomized, double blind, placebo controlled crossover pilot study. The participants will also perform morning typical behaviors such as arousal from sleep, change in posture (getting out of bed) and mild intensity physical activity; identical to the stressors encountered in everyday life. This pilot study is in healthy middle aged adults without a history of CV disease.

Participants will spend two nights in an inpatient hospital suite at Hatfield Research Center. Upon awakening in the morning, they will either ingest Vitamin C or placebo in a randomized order. This will be followed by moderate intensity exercise, recovery, and discharge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Normal weight or overweight but not obese (18.5<BMI<33 kg/m2)

Exclusion Criteria:

* History of smoking/tobacco use
* Current prescription/non-prescription medications or drugs of abuse
* Acute, chronic, or debilitating medical conditions
* History of working irregular day and night hours, regular night work, or rotating shift work for the six months prior to the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Vascular Endothelial Function | Approximately three months
  Vascular endothelial function will be measured as flow-mediated dilation (FMD). We will measure brachial artery FMD immediately upon awakening in a constant posture following an overnight fast using the standard guidelines and protocol.
Oxidative stress | Approximately three months
  Oxidative stress will be measured as malondialdehyde (MDA) adducts from Ethylenediaminetetraacetic acid (EDTA) plasma. Higher values may indicate increased oxidative stress.
Plasma Vitamin C and Tetrahydrobiopterin | Approximately three months
  We will measure Vitamin C levels in the plasma to ensure that the levels are increased after supplementation, and to control for baseline levels. We will measure tetrahydrobiopterin (BH4) from plasma to test if levels are increased upon administration of Vitamin C.

SECONDARY OUTCOMES:
Platelet aggregation | Approximately three months
  Platelet aggregation will be measured using Chronolog 560 VS Platelet aggregometer as an indicator of how well blood clots or clumps together. Higher values may indicate increased cardiovascular risk.
Plasminogen activator inhibitor -1 | Approximately three months
  Plasminogen activator inhibitor-1 (PAI-1) will be measured from plasma as a blood inflammatory marker. Higher values may indicate increased cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh S Thosar, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No